CLINICAL TRIAL: NCT00615446
Title: A Phase 1 Study Of SU011248 And Gemcitabine In Patients With Advanced Solid Tumors
Brief Title: A Study To Find The Best Doses Of SU011248 And Gemcitabine When Given Together To Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181041
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Solid Tumors
Keywords: solid tumor malignancy, SU011248, sunitinib, neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Sunitinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: SU011248; Gemcitabine

INTERVENTIONS:
Drug: SU011248; Gemcitabine — Dose finding study using SU011248 (sunitinib) daily by oral capsule in 4/2 (administered for 4 out of every 6 weeks) or 2/1 (administered for 2 out of every 3 weeks) schedule with gemcitabine administered on Days 1, 8, 22 and 29 on Schedule 4/2 and Days 1 and 8 on Schedule 2/1 until progression or unacceptable toxicity
  Other Names: Sutent, sunitinib, SU11248, Gemzar

SUMMARY:
This study assesses the maximum tolerated dose, overall safety and antitumor activity of SU011248 in combination with gemcitabine in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of a solid cancer which is not responsive to standard therapy or for which no standard therapy exists
* Patient has good performance status (ECOG 0 or 1)

Exclusion Criteria:

* Prior treatment with either gemcitabine or SU011248
* Hypertension that cannot be controlled by medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximally tolerated dose of SU011248 (dosed on Schedule 4/2 or 2/1) when given in combination with gemcitabine | From screening until at least 28 days beyond discontinuation of study treatment

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of SU011248 and gemcitabine when these drugs are co-administered | From screening until at least 28 days beyond discontinuation of study treatment
To preliminarily assess the antitumor activity of SU011248 and gemcitabine in patients with measurable disease | From screening until at least 28 days beyond discontinuation of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Michaelson MD, Zhu AX, Ryan DP, McDermott DF, Shapiro GI, Tye L, Chen I, Stephenson P, Patyna S, Ruiz-Garcia A, Schwarzberg AB. Sunitinib in combination with gemcitabine for advanced solid tumours: a phase I dose-finding study. Br J Cancer. 2013 Apr 16;108(7):1393-401. doi: 10.1038/bjc.2013.96. Epub 2013 Mar 19. PMID 23511559
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181041&StudyName=A%20Study%20To%20Find%20The%20Best%20Doses%20Of%20SU011248%20And%20Gemcitabine%20When%20Given%20Together%20To%20Patients%20With%20Advanced%20Solid%20Tumors